CLINICAL TRIAL: NCT01504867
Title: LIPS-A: Lung Injury Prevention Study With Aspirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Montefiore Medical Center (Other); Vanderbilt University Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Daryl J. Kor, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-004856; U01HL108712-01 (NIH); KL2RR024151 (NIH); K23HL112855 (NIH); UL1TR000433 (NIH)
Record Dates: First submitted 2012-01-03; First posted 2012-01-06 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; ARDS; ALI; aspirin; prevention
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): This arm received a 325mg loading dose of aspirin on study day one, followed by 81mg of aspirin on days 2-7.
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): This group received matching lactose powder filled capsules on days 1-7.
  Interventions: Drug: Lactose powder

INTERVENTIONS:
Drug: Aspirin — 325mg loading dose once on study day 1, followed by 81mg dose once daily on study days 2-7. Administered by mouth or down nasal gastric tube.
  Arms: Aspirin
Drug: Lactose powder — Matching lactose powder filled capsules will be administered on days 1-7.
  Arms: Placebo

SUMMARY:
The primary hypothesis was that early aspirin administration will decrease the rate of developing acute lung injury during the first 7 days after presentation to the hospital.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) remains a life-threatening critical care syndrome characterized by alveolar-capillary membrane injury and hypoxemic respiratory failure. The median time to onset of ARDS is 2 days after hospital presentation. Therefore, the period between hospital presentation and the development of ARDS presents a brief window of opportunity for ARDS prevention.

This was a multicenter, double-blind, placebo-controlled, parallel-group, Phase 2b, randomized clinical trial. Development of ARDS was defined by Berlin criteria (modified to require invasive mechanical ventilation) within 7 days of hospital admission. The first dose of study drug or placebo was administered within 24 hours after presentation to the hospital. Important co-interventions were standardized across sites using a web-based tool, Checklist for Lung Injury Prevention. Study participants were screened daily for receipt of mechanical ventilation and determination of the partial pressure of arterial oxygen (PaO2) or oxygen saturation to fraction of inspired oxygen ratio (SpO2:FIO2). If the participant's SpO2:FIO2 ratio was consistently below 315, hypoxemia was confirmed with measurement of arterial blood gas. Chest radiographs for all intubated patients with a SpO2:FIO2 of 300 or less were independently reviewed by both site investigator and a member of the trial's executive committee. Study participants who died or were discharged from the hospital before day 7 without meeting criteria for ARDS were adjudicated as not having ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18) admitted to the hospital through the emergency department (ED)
* At high risk of developing acute lung injury (ALI) Lung Injury Prediction Score (LIPS) greater than or equal to 4

Exclusion Criteria:

* Anti-platelet therapy on admission or within 7 days prior to admission
* Presented to outside hospital ED > 12 hrs before arrival at site's facility
* Inability to obtain consent within 12 hours of hospital presentation
* Admitted for elective surgery
* Acute lung injury prior to randomization
* Receiving mechanical ventilation through a tracheostomy tube prior to current hospital admission (patient who is ventilator dependent)
* Presence of bilateral pulmonary infiltrates on admission if he or she has a history of bilateral pulmonary infiltrates (as evidenced by previous x-rays) that can reasonably explain the current degree of pulmonary infiltrates present.
* Presentation due to pure heart failure and no other known risk factors for ALI.
* Allergy to aspirin or non steroidal anti inflammatory drugs (NSAIDs)
* Bleeding disorder
* Suspected active bleeding or judged to be at high risk for bleeding
* Active peptic ulcer disease (within past 6 months)
* Severe chronic liver disease
* Inability to administer the study drug
* Expected hospital stay < 48 hours
* Admitted for comfort or hospice care
* Patient, surrogate or physician not committed to full support. (Exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
* Not anticipated to survive > 48 hours
* Previously enrolled in this trial
* Enrolled in a concomitant intervention trial
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Kor, MD, Principal Investigator — Mayo Clinic
Locations (16):
- United States (16):
  - Stanford Univeristy, Stanford, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - University of Florida, Gainsville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Louisville Medical Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kor DJ, Carter RE, Park PK, Festic E, Banner-Goodspeed VM, Hinds R, Talmor D, Gajic O, Ware LB, Gong MN; US Critical Illness and Injury Trials Group: Lung Injury Prevention with Aspirin Study Group (USCIITG: LIPS-A). Effect of Aspirin on Development of ARDS in At-Risk Patients Presenting to the Emergency Department: The LIPS-A Randomized Clinical Trial. JAMA. 2016 Jun 14;315(22):2406-14. doi: 10.1001/jama.2016.6330. PMID 27179988
- [Derived] Abdulnour RE, Gunderson T, Barkas I, Timmons JY, Barnig C, Gong M, Kor DJ, Gajic O, Talmor D, Carter RE, Levy BD. Early Intravascular Events Are Associated with Development of Acute Respiratory Distress Syndrome. A Substudy of the LIPS-A Clinical Trial. Am J Respir Crit Care Med. 2018 Jun 15;197(12):1575-1585. doi: 10.1164/rccm.201712-2530OC. PMID 29782179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 1/2/2012 and 11/17/2014 at multiple US academic hospitals.
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 202 | 198
Completed | 195 | 195
Not Completed | 7 | 3
Not completed — Inclusion criteria not met | 2 | 2
Not completed — Consent revoked | 5 | 1

BASELINE CHARACTERISTICS:
Population: 400 subjects were randomized, and 10 subjects were excluded, leaving 390 in the final modified intention-to-treat analysis cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 195 | 195 | 390
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57.0 [44.0 to 67.0] | 57.0 [47.0 to 68.0] | 57 [45 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 99 | 187
  Male | 107 | 96 | 203
Region of Enrollment [Number; unit: participants]
  United States | 195 | 195 | 390

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Acute Respiratory Distress Syndrome (ARDS) Within 7 Days
Description: ARDS was defined by Berlin criteria (modified to require invasive mechanical ventilation) within 7 days of hospital admission.
Time Frame: Within seven days from hospital presentation
Population: Intention-to-Treat
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
participants | 20 | 17
Statistical Analysis 1: Comparison: Aspirin vs Placebo; The primary outcome significance level was adjusted for multiple testing associated with the interim analysis. Its significance level is 92.6%; Test type: Superiority or Other; p = 0.53, Wald; This was a large sample (Wald) test estimated using a conditional logistic regression model with site as a stratification variable

2. Secondary Outcome: Hospital Mortality
Time Frame: 28 days
Population: Intention-to-Treat
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
participants | 14 | 14
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p > 0.99, Chi-squared

3. Secondary Outcome: Number of Participants With ARDS or Mortality Within 7 Days
Time Frame: within 7 days
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
participants | 27 | 21
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 0.36, Chi-squared

4. Secondary Outcome: Number of Subjects With Mechanical Ventilation at Any Time During Hospitalization
Time Frame: approximately 7 days
Population: Intention-to-Treat
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
participants | 51 | 41
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 0.23, Chi-squared

5. Secondary Outcome: Mean Number of Days Participants Were Ventilator-Free To Day 28
Time Frame: baseline, Day 28
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
days | 24.9 (7.4) | 25.2 (7.0)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Subjects Admitted to Intensive Care Unit (ICU)
Time Frame: 7 days
Population: Intention-to-Treat
Measure: Number; unit: participants
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
participants | 115 | 98
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 0.08, Chi-squared

7. Secondary Outcome: Mean Hospital Length of Stay
Time Frame: approximately 7 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 195 | 195
days | 8.8 (10.3) | 9.0 (9.9)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Aspirin | Placebo
Serious Adverse Events (participants affected / at risk) | 4/195 | 8/195
Other Adverse Events (participants affected / at risk) | 13/195 | 5/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=195) | Placebo (N=195)
Bleeding Stress Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia due to Upper GI Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia/Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 0 (0) | 1 (2)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=195) | Placebo (N=195)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cerebral Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Elevated Blood Pressure (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Mild Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
Nose Bleed (Vascular disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal Bleeding (Renal and urinary disorders) | 1 (1) | 0 (0)
Right Hip Resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Urosepsis (Renal and urinary disorders) | 1 (1) | 0 (0)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Renal Failure Requiring Dialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No